CLINICAL TRIAL: NCT06212895
Title: Attitude and Expectations of Patients Regarding Exercise and Physical Activity as a Therapeutic Option in an Orthopedic Outpatient Clinic - A Cross-Sectional-Trial
Brief Title: Expectations of Patients Regarding Exercise in an Outpatient Clinic
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Regensburg (Other)
Collaborators: OCS Straubing (Unknown)
Responsible Party: Principal Investigator, Thomas Okon, MD, University of Regensburg
Other Study IDs: 23-3534-101
Record Dates: First submitted 2023-12-08; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Communcation; Physical Activity; Prescription
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — A survey is handled out at the patient registration. Patients can fill it out during waiting for their appointment. The physician, who treats the patients is not aware aout the filling status or content. The Survy will not influence the treatment.
  The Survey consists of 3 parts: patients attidude and expectations, and questionnaire about their usual physical activity and the validated Expectation Treatment Score.

SUMMARY:
Exercise and physical activity are recommended in many clinical guidelines in orthopdeci diseases. Costs, time, doctor-patient-communication and the type of prescription are possible limitations of prescribing exercise as a therapy. It is essential to know the expactiations and attitude of the patients for an accurate, patient-centered, prescription. This trial aims to reveal patients point of view and attitude.

ELIGIBILITY:
Inclusion Criteria:

* patient presented the first time in the outpatient study with an issue

Exclusion Criteria:

* language barrier
* cognitive impairment which could lead to missunderstadning of the survey

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes patients, which present themself for the first time in this outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Attitude of patients regarding exercise and physical activity as a therapeutic option | July 2024
  - measured via Likert Scale. The attitude is derived from multiple questions in a survey ("In my opinion, exercise is as effective as an intervention/operation", etc.

SECONDARY OUTCOMES:
influencing factors of patients attitude | July 2024
  descriptive statistics and regression analysis regarding patient characteristics, measured via surveys (social background, highest graduation; positive experience with exercise as therapeutic option; age in years, bodyweight (kg), kind of orthopedic disease (tendinopathy, arthrosis, disc herniation (nominal categories)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Epidemiology and Preventive Medicine, Division of Medical Sociology, University of Regensburg, Regensburg, Germany